CLINICAL TRIAL: NCT02090062
Title: Difference in H. Pylori Infection Rate of EGC Patients Before and After Endoscopic Resection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjxhnk2014
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Early Gastric Cancer
Keywords: endoscopic resection; H. pylori infection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All the lesions will be removed endoscopically or surgically and examine histologically by an independent gastrointestinal pathologist.
  Each biospecimen after ER will be detected H pylori infection status.
Oversight: Data Monitoring Committee: No

SUMMARY:
Parts of patients are diagnosed as H. pylori -negative before ER, whereas the specimens become H. pylori-positive after ER, which may have a role in the recurrence of EGC. Our study aims to determine the difference in H. pylori infection rate of EGC patients before and after ER , and discuss the causes leading to the difference, which can provide references for improving the diagnostic accuracy of H. pylori infection and reducing EGC's recurrence rate.

DETAILED DESCRIPTION:
Gastric cancer is the fourth most commonly diagnosed cancer in the world and the second leading cause of cancer-related deaths. Nowadays, endoscopic resection（ER） is widely accepted as the primary treatment for early gastric cancer (EGC) without lymph node metastasis，which includes endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD).However, recurrence rate after endoscopic resection for EGC still achieves 6.7%-14%. However, there is no comparative analysis about H. pylori infection rate before and after ER yet.

ELIGIBILITY:
Inclusion Criteria:

* high grade dysplasia(HGD) and EGC patients treated by endoscopic resection(including EMR and ESD) in Ren Ji hospital

Exclusion Criteria:

* Suspect of advanced gastric cancer
* Lesions with light grade dysplasia
* History of gastric surgery
* Poor gastrointestinal preparation
* Patients under unsuitable conditions for examination or treatment, such as acute upper gastrointestinal bleeding, noncorrectable coagulopathy, severe systemic disease, etc

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with early gastric lesions
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
difference in H. pylori infection rate before and after ER | in two weeks after endoscopic resection
  Information on the H pylori infection status before ER will be collected from the medical records of each patient. A positive result on at least one rapid urease test, urease breath test or Giemsa staining is deemed to be indicative of H pylori infection .Each specimen after ER will be detected H pylori infection status in two weeks. Then we analyze the difference in H. pylori infection rate before and after ER.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Li, MD.Ph.D, Principal Investigator — Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai,China,Shanghai Institute of Digestive Disease, Shanghai,China